CLINICAL TRIAL: NCT04917302
Title: Combination of NMDA-enhancing and Anti-inflammatory Treatments for Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH108-REC1-178
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA; Inflammation
MeSH Terms: conditions — Schizophrenia; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE plus Anti-inflammatory Agent (AIFA) (Experimental): An NMDA enhancer plus a drug with anti-inflammatory property
  Interventions: Drug: NMDAE plus AIFA
- NMDAE plus Placebo (Placebo Comparator): An NMDA enhancer plus Placebo
  Interventions: Drug: NMDAE plus Placebo Cap

INTERVENTIONS:
Drug: NMDAE plus AIFA — Use of an NMDA enhancer plus a drug with anti-inflammatory property for the treatment of schizophrenia.
  Arms: NMDAE plus Anti-inflammatory Agent (AIFA)
Drug: NMDAE plus Placebo Cap — Use of an NMDA enhancer plus placebo as a comparator
  Arms: NMDAE plus Placebo

SUMMARY:
Previous studies found that some NMDA-enhancing agents were able to improve clinical symptoms of patients with chronic schizophrenia. In addition, several drugs with anti-inflammatory properties have been tested in clinical trials for the treatment of schizophrenia too. Whether combined treatment of an NMDA-enhancing agent and a drug with anti-inflammatory property can be better than an NMDA-enhancing agent alone deserves study.

DETAILED DESCRIPTION:
Several lines of evidence suggest that both NMDA and inflammatory hypotheses have been implicated in schizophrenia. Previous studies found that some NMDA-enhancing agents were able to augment efficacy of antipsychotics in the treatment of chronic schizophrenia. In addition, several drugs with anti-inflammatory properties have been tested in clinical trials for the treatment of schizophrenia too. Whether a drug with anti-inflammatory property can strengthen the efficacy of an NMDA-enhancer (NMDAE) in the treatment of schizophrenia remains unknow. Therefore, this study aims to compare NMDAE plus a drug with anti-inflammatory property and NMDAE plus placebo in the treatment of schizophrenia. The subjects are the patients with treatment-resistant schizophrenia who have responded poorly to two or more kinds of antipsychotics treatment. They keep their original treatment and are randomly, double-blindly assigned into two treatment groups for 12 weeks: (1) NMDAE plus Anti-inflammatory Agent (AIFA), or (2) NMDAE plus placebo. Clinical performances and side effects are measured at weeks 0, 2, 4, 6, 9, and 12. Cognitive functions are assessed at baseline and at endpoint of treatment by a battery of tests. The efficacies of NMDAE plus AIFA and NMDAE plus placebo will be compared.

Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-5 (American Psychiatric Association) diagnosis of schizophrenia
* Are resistant to adequate treatments of at least two antipsychotics
* Remain symptomatic but without clinically significant fluctuation, while their antipsychotic doses are unchanged for at least 3 months and will be maintained during the period of the 12-week trial
* PANSS total score ≥ 70
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* DSM-5 diagnosis of intellectual disability or substance (including alcohol) use disorder
* History of epilepsy, head trauma, stroke, or serious medical or central nervous system diseases (other than schizophrenia) which may interfere with the study
* Clinically significant laboratory screening tests (including blood routine, biochemical tests)
* Pregnancy or lactation
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of Positive and Negative Syndrome Scale (PANSS) | week 0, 2, 4, 6, 9, 12]
  Assessment of overall symptoms. Minimum value: 30, maximum value:210, the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change of scales for the Assessment of Negative Symptoms (SANS) total score | 0, 2, 4, 6, 9, 12
  Assessment of negative symptoms. Minimum value: 0, maximum value:100, the higher scores mean a worse outcome.
Positive subscale, Negative subscales, and General Psychopathology subscale of PANSS | week 0, 2, 4, 6, 9, 12
  PANSS-positive: Assessment of positive symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
  PANSS-negative: Assessment of negative symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
  PANSS-general psychopathology: Assessment of general psychopathology. Minimum value: 16, maximum value:112, the higher scores mean a worse outcome
Clinical Global Impression | week 0, 2, 4, 6, 9, 12
  Assessment of general impression. Minimum value: 1, maximum value:7, the higher scores mean a worse outcome.
Global Assessment of Functioning | week 0, 2, 4, 6, 9, 12
  Assessment of social, occupational, and psychological function. Minimum value: 1, maximum value:100, the higher scores mean better function.
Hamilton Rating Scale for Depression | week 0, 2, 4, 6, 9, 12
  Assessment of depressive symptoms. Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.
Quality of Life Scale | week 0, 2, 4, 6, 9, 12
  Assessment of life quality. Minimum value: 0, maximum value:126, the higher scores mean a better outcome.
Cognitive function | Week 0, 12
  The measure is the composite from multiple measures.
  Ten cognitive tests for assessment of 7 cognitive domains:
  1. speed of processing (assessed by 3 tests: Category Fluency, Trail Marking A, WAIS-III Digit Symbol-Coding);
  2. sustained attention (Continuous Performance Test);
  3. working memory: verbal (digit span) and nonverbal (spatial span);
  4. verbal learning and memory (WMS-III, word listing);
  5. visual learning and memory (WMS-III, visual reproduction);
  6. reasoning and problem solving (WISC-III, Maze);
  7. social cognition (the Mayer-Salovey-Caruso Emotional Intelligence Test [MSCEIT] Version 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan